CLINICAL TRIAL: NCT03899090
Title: Investigating Floatation-REST as a Novel Technique for Reducing Anxiety and Depression
Brief Title: Floatation-REST (Reduced Environmental Stimulation Therapy) for Anxiety and Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Float R34; R34AT009889 (NIH)
Record Dates: First submitted 2019-03-04; First posted 2019-04-02 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Generalized Anxiety Disorder; Social Anxiety Disorder; Panic Disorder; Agoraphobia; Posttraumatic Stress Disorder; Major Depressive Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder; Phobia, Social; Panic Disorder; Agoraphobia; Stress Disorders, Post-Traumatic; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of three arms:
  1. floating supine in a pool for a prescribed amount of time (6 total sessions, 1 hour/session, 1 session/week)
  2. floating supine in a zero-gravity chair for a prescribed amount of time (6 total sessions, 1 hour/session, 1 session/week)
  3. floating supine in a pool for a preferred amount of time (6 total sessions, up to 2 hours/session, as frequently as they prefer within a 12-week period with a minimum of 24 hours between sessions)
Who Masked: Participant, Investigator
Masking Description: The investigator and participant are masked to study arm until after the participant completes their baseline session, at which point they are randomized using a sealed envelope.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Float Pool (Experimental): Floating supine in a pool for a prescribed amount of time (6 total sessions, 1 hour/session, 1 session/week)
  Interventions: Behavioral: Float pool
- Float Chair (Active Comparator): Floating supine in a zero-gravity chair for a prescribed amount of time (6 total sessions, 1 hour/session, 1 session/week)
  Interventions: Behavioral: Float chair
- Float Pool Preferred (Experimental): Floating supine in a pool for a preferred amount of time (6 total sessions, up to 2 hours/session, as frequently as they prefer within a 12-week period with a minimum of 24 hours between sessions)
  Interventions: Behavioral: Float pool

INTERVENTIONS:
Behavioral: Float pool — Subject floats supine in a pool of water saturated with Epsom salt in an environment which minimizes stimulation of the nervous system, including reduced light, sound, and pressure on the spinal cord.
  Arms: Float Pool; Float Pool Preferred
Behavioral: Float chair — Subject floats supine in a zero-gravity chair in an environment which minimizes stimulation of the nervous system, including reduced light, sound, and pressure on the spinal cord.
  Arms: Float Chair

SUMMARY:
This early-stage trial aims to examine the feasibility, tolerability, and safety of Floatation-REST (Reduced Environmental Stimulation Therapy) or an active comparison condition in 75 participants with clinical anxiety and depression.

DETAILED DESCRIPTION:
Anxiety and depression are the two most common psychiatric conditions, affecting over a quarter of the population, and representing the leading cause of disability, worldwide. More than three-quarters of patients never receive treatment, and recent meta-analyses and large-scale clinical trials suggest that only about half of patients improve with treatment, with substantially poorer outcomes and adherence in patients with comorbid anxiety and depression. Given the insufficient treatment response and adherence to currently available therapies, it is important to explore novel ways of helping patients with anxiety and depression. Floatation-REST (Reduced Environmental Stimulation Therapy) is a relatively unexplored mind-body intervention for naturally reducing physiological stress by attenuating exteroceptive sensory input to the nervous system through the act of floating supine in a pool of water saturated with Epsom salt (magnesium sulfate). Over the past decade, floating has witnessed a rapid rise in popularity, with hundreds of recreational float centers opening across America. Despite the surge in public interest and consumption, there has been little research investigation Floatation-REST, especially in clinical populations. The investigators recently completed several pilot studies in patients with comorbid anxiety and depression showing that a single float session was capable of inducing a large short-term anxiolytic and antidepressant response accompanied by a substantial improvement in mood and subjective well-being. This proposal aims to follow-up on these promising preliminary findings by investigating the feasibility, tolerability, and safety of undergoing multiple sessions of Floatation-REST or an active comparison condition in 75 participants with clinical anxiety and depression. A subset of these participants will have the opportunity to select their preference with regard to float duration and frequency, providing important information for optimizing the "dose" in future trials. Since this study is aimed at examining feasibility, tolerability, and safety, the primary endpoint is adherence (as a proxy of feasibility), and the secondary outcome measures are dropout rate (as a proxy for tolerability) and adverse effects (as a proxy for safety). An exploratory aim examines the magnitude and duration of the anxiolytic and antidepressant effects of Floatation-REST at both short-term (up to 48 hours) and long-term (up to 6 months) intervals, providing an initial indication for whether any beneficial effects are sustained beyond the float experience. The results of this early phase clinical trials will help optimize the design of a future efficacy study exploring the long-term effects of Floatation-REST.

ELIGIBILITY:
Inclusion Criteria:

1. High level of acute anxiety (OASIS score ≥ 6)
2. High anxiety sensitivity (ASI-3 total score ≥ 24)
3. If taking medication or receiving psychotherapy, must be stably undergoing treatment prior to participation (defined as having taken the medication or been in therapy for 8 weeks or longer). If taking a benzodiazepine or opioid, must be willing to abstain within 24 hours of a float session (daily users will be excluded from the study).
4. No prior Floatation-REST experience or a minimum of 1 year since previous float session
5. Seeking treatment for their anxiety/depression and willing to complete the study

Exclusion Criteria:

1. History of Bipolar Disorder, Schizophrenia spectrum or other psychotic disorders
2. Current Eating Disorder (anorexia/bulimia nervosa)
3. Current Substance Use Disorder ≥ moderate. Tobacco and Caffeine Use is allowed. Must be willing to abstain from all other substances within 24 hours of a float session.
4. Active suicidality with plan/intent
5. History of a neurological condition (e.g., epilepsy) or any other medical condition that could interfere with the protocol
6. Any skin conditions or open wounds that could cause pain when exposed to saltwater
7. Uncomfortable being in water
8. Positive pregnancy test
9. Acutely intoxicated day of floating (determined via positive urine drug screen or breathalyzer)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Adherence | Over 6-9 week period of intervention (up to 12 weeks for preferred pool arm)
  As a proxy of feasibility, adherence for each subject = (# of sessions completed)/6.
  All subjects (in all arms of the study) are given up to 3 opportunities to reschedule missed appointments, after which they are withdrawn from the study.

SECONDARY OUTCOMES:
Dropout rate | Over 6-9 week period of intervention (up to 12 weeks for preferred pool arm)
  As a proxy for tolerability, dropout rate for each arm = (# of subjects who are withdrawn from the study)/25.
  All subjects (in all arms of the study) are given up to 3 opportunities to reschedule missed appointments, after which they are withdrawn from the study.
Adverse effects | Over 6-9 week period of intervention (up to 12 weeks for preferred pool arm)
  As a proxy of safety, adverse effects for each subject = # of instances during the study when a subject reports elevations above mild for any negative effects on the side effect checklist (administered after each float session)
Psychological Distress on the Brief Symptom Inventory-18 | Through study completion, an average of 6 months after the final float session
  Total Score on the Brief Symptom Inventory-18 [Average change pre to post-intervention]
Anxiety on the Brief Symptom Inventory-18 | Through study completion, an average of 6 months after the final float session
  Anxiety subscale [Average change pre to post-intervention]
Depression on the Brief Symptom Inventory-18 | Through study completion, an average of 6 months after the final float session
  Depression subscale [Average change pre to post-intervention]
Somatization on the Brief Symptom Inventory-18 | Through study completion, an average of 6 months after the final float session
  Somatization subscale [Average change pre to post-intervention]
Anxiety on the clinician-rated Hamilton Anxiety Rating Scale (HAM-A) | Through study completion, an average of 6 months after the final float session
  Total score [Average change pre to post-intervention]
Depression on the clinician-rated Montgomery Åsberg Rating Scale (MADRS) | Through study completion, an average of 6 months after the final float session
  Total score [Average change pre to post-intervention]
Disability on the Sheehan Disability Scale | Through study completion, an average of 6 months after the final float session
  Total score [Average change pre to post-intervention]
Anxiety remission | An average of 6 weeks after the final float session
  Percent of individuals by condition (chair, pool, pool-preferred) who have a HAM-A score of ≤ 7
Anxiety responder | Through study completion, an average of 6 months after the final float session
  Percent of individuals by condition (chair, pool, pool-preferred) who show a 50% reduction on HAM-A or Overall Anxiety Severity and Impairment Scale (OASIS)
Depression remission | An average of 6 weeks after the final float session
  Percent of individuals by condition (chair, pool, pool-preferred) who have a MADRS score of ≤ 9
Depression responder | Through study completion, an average of 6 months after the final float session
  Percent of individuals by condition (chair, pool, pool-preferred) who show a 50% reduction on MADRS or Patient Health Questionnaire-9 (PHQ-9)
Depression on the Patient Health Questionnaire-9 (PHQ-9) | Through study completion, an average of 6 months after the final float session
  Total score [Average change pre to post-intervention]
Anxiety on the Overall Anxiety Severity and Impairment Scale (OASIS) | Through study completion, an average of 6 months after the final float session
  Total score [Average change pre to post-intervention]
Anxiety Sensitivity on the Anxiety Sensitivity Index-3R (ASI-3R) | Through study completion, an average of 6 months after the final float session
  Total score [Average change pre to post-intervention]
Positive Affect on the Positive and Negative Affect Schedule-X (PANAS-X) | Through completion of the final float session
  Average of Positive Affect rating change scores from pre-to-post float across all six floats for each condition (chair, pool, pool-preferred)
Negative Affect on the Positive and Negative Affect Schedule-X (PANAS-X) | Through completion of the final float session
  Average of Negative Affect rating change scores from pre-to-post float across all six floats for each condition (chair, pool, pool-preferred)
Serenity on the Positive and Negative Affect Schedule-X (PANAS-X) | Through completion of the final float session
  Average of Serenity rating change scores from pre-to-post float across all six floats for each condition (chair, pool, pool-preferred)
State Anxiety on the State Trait Anxiety Inventory (STAI) | Through completion of the final float session
  Average of STAI State Anxiety rating change scores from pre-to-post float across all six floats for each condition (chair, pool, pool-preferred)
Muscle Tension rating on the Visual Analog Scale (VAS) | Through completion of the final float session
  Average of VAS muscle tension rating change scores from pre-to-post float all six floats for each condition (chair, pool, pool-preferred)
Pain on the Wong-Baker Pain Scale (WBPS) | Through completion of the final float session
  Average of WBPS rating change from pre-to-post float across all six floats for each condition
Trait Anxiety on the State Trait Anxiety Inventory | Through study completion, an average of 6 months after the final float session
  Average of STAI Trait Anxiety rating change scores from pre-to-post float across all six floats for each condition (chair, pool, pool-preferred)
Cardiac interoceptive accuracy | Through completion of the final float session
  Average of Beat-to-squeeze consistency on cardiac interoception task
Heartbeat perception rating | Through completion of the final float session
  Average of heartbeat intensity, task difficulty, and task accuracy ratings

OTHER OUTCOMES:
Blood concentration (pg/mL) of proinflammatory cytokines (IFN-γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13, and TNF-α) | Blood samples collected at 3 time points: beginning of intervention (baseline), end of intervention (6-9 weeks after baseline), and at 6-week follow-up (12-15 weeks after baseline).
  At each time point, 10 cytokines will be measured in the blood as well as in response to a potent immune stressor (endotoxin)

CONTACTS AND LOCATIONS:
Overall Officials: Sahib Khalsa, MD, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the study results will be deidentified and shared with interested investigators using an online link
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal

REFERENCES:
- [Derived] Garland MM, Wilson R, Thompson WK, Stein MB, Paulus MP, Feinstein JS, Khalsa SS. A randomized controlled safety and feasibility trial of floatation-REST in anxious and depressed individuals. PLoS One. 2024 Jun 6;19(6):e0286899. doi: 10.1371/journal.pone.0286899. eCollection 2024. PMID 38843272
- [Derived] Garland MM, Wilson R, Thompson WK, Stein MB, Paulus MP, Feinstein JS, Khalsa SS. A randomized controlled safety and feasibility trial of floatation-REST in anxious and depressed individuals. medRxiv [Preprint]. 2023 Jun 8:2023.05.27.23290633. doi: 10.1101/2023.05.27.23290633. PMID 37333146